CLINICAL TRIAL: NCT06741787
Title: Microbial Characterization in Patients With Allergic Rhinitis Before and After Sublingual Immunotherapy Spray
Brief Title: Microbial Study of Sublingual Immunotherapy Spray in Patients With Allergic Rhinitis
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-SR-961
Record Dates: First submitted 2024-01-22; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — elbow venous blood: 2ml, feces: 5ml, saliva:2ml, tonsil microorganism:2ml, nasal exfoliated cells:2ml, nasal microorganism:2ml.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients desensitized by sublingual spray: Oraltekzc®️(Canis familiari), Oraltek®️(Felis domesticus), Oraltek®️(Alternaria alternata), dosage form: sublingual spray.
  Interventions: Drug: Patients desensitized by sublingual spray

INTERVENTIONS:
Drug: Patients desensitized by sublingual spray — Drug: Oraltekzc®️(Canis familiari), Oraltek®️(Felis domesticus), Oraltek®️(Alternaria alternata), dosage form: sublingual spray.

SUMMARY:
The incidence of allergic rhinitis (AR) in Chinese adults was reported to be as high as 24.1% and 16.8% in children. The current symptomatic treatment has the disadvantage of poor efficacy and cannot change the natural course of the disease. Allergen immunotherapy (AIT) is the only causative treatment approved by the WHO, bringing a new option to patients with allergic diseases. The quality of allergen preparations is critical to the diagnosis and treatment of the disease, emphasizing the need for standardized preparations, and AIT treatment in the early stages of the disease may change the long-term progression of the disease. Recent studies have reported that the microbiome of patients with different efficacy of desensitization therapy is different and may be correlated with the clinical symptoms of patients, but no prospective studies have been reported.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-65 years).
* Patients with canis familiari/felis domesticus/alternaria alternata allergic rhinitis were diagnosed based on clinical history and positive dust mite sensitization tests (skin prick test and/or specific IgE).
* Patients who visited the Department of Otolaryngology of the First Affiliated Hospital of Nanjing Medical University and selected sublingual spray desensitization.

Exclusion Criteria:

* Patients who refused to accept specimen and questionnaire collection.
* Patients who had nasal diseases other than allergic rhinitis, such as nasal papilloma and nasal malignant tumor.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with allergic rhinitis in the Department of Otolaryngology of the First Affiliated Hospital of Nanjing Medical University and selected sublingual spray desensitization.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | 2024.2-2026.7
  Patients were scored by questionnaire before and after treatment, and the change in score before and after treatment was the primary outcome measure
Visual analogue scale (VAS) | 2024.2-2026.7
  Patients were scored by questionnaire before and after treatment, and the change in score before and after treatment was the primary outcome measure. Range: 0-10. Higher scores reflect more pain and severity.
Total Nasal Symptom Score (TNSS) | 2024.2-2026.7
  It includes four common nasal symptoms: itching, nasal congestion, sneezing and runny nose. These four symptoms are scored using a "four-point scale," in which the severity of each symptom is rated from 0 to 3. The total score for the entire TNSS score is the sum of the four symptom scores, which range from 0 to 12.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Cheng, PhD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China